CLINICAL TRIAL: NCT00000556
Title: Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 100
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2005-11

CONDITIONS: Arrhythmia; Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases | interventions — Amiodarone; Sotalol; Propafenone; Flecainide; Quinidine; Moricizine; Disopyramide; Procainamide; Adrenergic beta-Antagonists; Verapamil; Diltiazem; Digoxin; Catheter Ablation; Pacemaker, Artificial

INTERVENTIONS:
Drug: amiodarone
Drug: sotalol
Drug: propafenone
Drug: flecainide
Drug: quinidine
Drug: moricizine
Drug: disopyramide
Drug: procainamide
Drug: adrenergic beta antagonists
Drug: verapamil
Drug: diltiazem
Drug: digoxin
Procedure: catheter ablation
Device: pacemaker, artificial

SUMMARY:
To compare two standard treatment strategies for atrial fibrillation: ventricular rate control and anticoagulation vs. rhythm control and anticoagulation.

DETAILED DESCRIPTION:
BACKGROUND:

Atrial fibrillation is an extremely common and increasingly prevalent cardiac arrhythmia, particularly in the elderly, and is an important risk factor for stroke. Management of atrial fibrillation remains controversial, and although antiarrhythmic drugs are widely used for this condition, clinical studies to support their use are meager. Management of atrial fibrillation has at least three components: restoration and maintenance of sinus rhythm; heart rate control when maintenance of sinus rhythm or when cardioversion is not attempted or impossible; and anticoagulation. The first component of management uses antiarrhythmic drugs and the second uses a different group of antiarrhythmic drugs and catheter ablation. The third is anticoagulant therapy for patients in whom normal sinus rhythm cannot be maintained or in whom cardioversion is not attempted.

The initiative was developed by staff of the Clinical Trials Branch and the NHLBI Working Group on Atrial Fibrillation which met in Bethesda in April, 1993. The initiative was given concept clearance by the February 1994 National Heart, Lung, and Blood Advisory Council. The Request for Proposals was released in May 1994.

DESIGN NARRATIVE:

A randomized multicenter trial. The trial enrolled only patients with atrial fibrillation who were at high risk for stroke, that is, over 65 years of age or less than 65 and with one or more other risk factors for stroke such as systemic hypertension, diabetes mellitus, congestive heart failure, transient ischemic attack, prior cerebral vascular accident. High risk patients were treated with the anticoagulant warfarin. Cardioversion (electrical or pharmacologic) might have been attempted before randomization, but if it was unsuccessful, the patient was excluded from further consideration for randomization. Normal sinus rhythm must have persisted for one hour or greater after cardioversion to qualify as successful cardioversion. Patients were randomly assigned to treatment groups which included maintenance of sinus rhythm or heart rate control. Both treatment groups had two steps.

In the maintenance of sinus rhythm group, the choice of drugs was left to the primary treating physician, to be chosen from amiodarone, sotalol, propafenone, flecainide, quinidine, moricizine, disopyramide, procainamide, and combinations of these drugs. Atrioventricular nodal blocking drugs were also administered unless contraindicated. The major substudy for AFFIRM randomized initial drug choice among amiodarone, sotalol, and class I drugs. Prior drugs which were ineffective or poorly tolerated were not repeated. There were various drug exclusions depending on the patient's condition. Patients in the maintenance of sinus rhythm group had multiple cardioversions as needed. If there was treatment failure or intolerance after two or more pharmacologic trials, patients were considered for innovative therapy in Step II. In Step II, two maintenance doses of amiodarone were included, a low dose of 100 to 200 mg/day and a normal dose of 300 to 400 mg/day. Each dose of amiodarone was considered to be a single drug trial, so that patients who received treatment with amiodarone at both dosage levels were considered to have had two drug trials. It was not mandatory that Step II therapies be applied in any individual patient. The following innovative Step II therapies were approved for use in the study: (1) ablation of an atrial focus in patients with type I atrial flutter, if it was clinically documented that the atrial flutter led to atrial fibrillation; (2) atrial pacing alone, with or without documented bradycardia; (3) atrial pacing and antiarrhythmic drugs, with either single site or multiple site atrial pacing; and (4) surgical maze or atrial isolation procedures at selected centers. Catheter-based ablative procedures, such as those attempting to mimic the maze procedure were not approved in this study. Implanted atrial cardioverter defibrillators were also not approved. All therapy was periodically reviewed and subject to modification by the Steering Committee with concurrence by the DSMB and the NHLBI. In the event that sinus rhythm was not maintainable by any treatment, patients crossed over to rate control and anticoagulation.

The heart rate control arm used heart rate as the therapeutic target, rather than dose of medications. Drug dosage was adjusted to achieve target heart rates. During atrial fibrillation, heart rate was assessed both at rest and during activity at each clinic visit. The pharmacologic therapies approved for use in this arm included: beta blockers, verapamil, diltiazem, digoxin, or combinations of these drugs . When Step I pharmacologic therapies failed after two or more drug trials, the treating physician could select an approved Step II innovative therapy. The two innovative therapies approved for use with the heart rate control arm were: (1) atrioventricular node modification by catheter ablation, with or without placement of a pacemaker, with or without continued drugs to slow atrioventricular node conduction, and (2) total atrioventricular junctional ablation and placement of a pacemaker.

The primary endpoint by which the two strategies were compared was total mortality, analyzed by intention-to-treat. Secondary endpoints were composite end points (total mortality, disabling intracranial bleed, stroke, disabling anoxic encephalopathy, cardiac arrest, major noncentral nervous system bleed, cost of therapy, and quality of life. Follow-up was a minimum of two years and an average of 3.5 years. Recruitment and intervention extended from November 1995 through October 1999 with 4,060 patients enrolled by 213 sites.

ELIGIBILITY:
Elderly men and women with atrial fibrillation and other risk factors for stroke.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1995-03; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: H. Greene — Statistics and Epidemiology Research Corporation (S.E.R.C.)

REFERENCES:
- [Background] Atrial fibrillation follow-up investigation of rhythm management -- the AFFIRM study design. The Planning and Steering Committees of the AFFIRM study for the NHLBI AFFIRM investigators. Am J Cardiol. 1997 May 1;79(9):1198-202. PMID 9164885
- [Background] Wyse DG. The AFFIRM trial: main trial and substudies-what can We expect? J Interv Card Electrophysiol. 2000 Jan;4 Suppl 1:171-6. doi: 10.1023/a:1009815606734. PMID 10590505
- [Background] Waldo AL. Management of atrial fibrillation: the need for AFFIRMative action. AFFIRM investigators. Atrial Fibrillation Follow-up Investigation of Rhythm Management. Am J Cardiol. 1999 Sep 15;84(6):698-700. doi: 10.1016/s0002-9149(99)00419-1. No abstract available. PMID 10498142
- [Background] AFFIRM Investigators. Atrial Fibrillation Follow-up Investigation of Rhythm Management. Baseline characteristics of patients with atrial fibrillation: the AFFIRM Study. Am Heart J. 2002 Jun;143(6):991-1001. doi: 10.1067/mhj.2002.122875. PMID 12075254
- [Background] Epstein AE, Vidaillet H, Greene HL, Curtis AB, Ellenbogen KA, Simmons T, Mickel M. Frequency of symptomatic atrial fibrillation in patients enrolled in the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. J Cardiovasc Electrophysiol. 2002 Jul;13(7):667-71. doi: 10.1046/j.1540-8167.2002.00667.x. PMID 12139289
- [Background] Wyse DG, Waldo AL, DiMarco JP, Domanski MJ, Rosenberg Y, Schron EB, Kellen JC, Greene HL, Mickel MC, Dalquist JE, Corley SD; Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) Investigators. A comparison of rate control and rhythm control in patients with atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1825-33. doi: 10.1056/NEJMoa021328. PMID 12466506
- [Background] AFFIRM First Antiarrhythmic Drug Substudy Investigators. Maintenance of sinus rhythm in patients with atrial fibrillation: an AFFIRM substudy of the first antiarrhythmic drug. J Am Coll Cardiol. 2003 Jul 2;42(1):20-9. doi: 10.1016/s0735-1097(03)00559-x. PMID 12849654
- [Background] Corley SD, Epstein AE, DiMarco JP, Domanski MJ, Geller N, Greene HL, Josephson RA, Kellen JC, Klein RC, Krahn AD, Mickel M, Mitchell LB, Nelson JD, Rosenberg Y, Schron E, Shemanski L, Waldo AL, Wyse DG; AFFIRM Investigators. Relationships between sinus rhythm, treatment, and survival in the Atrial Fibrillation Follow-Up Investigation of Rhythm Management (AFFIRM) Study. Circulation. 2004 Mar 30;109(12):1509-13. doi: 10.1161/01.CIR.0000121736.16643.11. Epub 2004 Mar 8. PMID 15007003
- [Background] Steinberg JS, Sadaniantz A, Kron J, Krahn A, Denny DM, Daubert J, Campbell WB, Havranek E, Murray K, Olshansky B, O'Neill G, Sami M, Schmidt S, Storm R, Zabalgoitia M, Miller J, Chandler M, Nasco EM, Greene HL. Analysis of cause-specific mortality in the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Circulation. 2004 Apr 27;109(16):1973-80. doi: 10.1161/01.CIR.0000118472.77237.FA. Epub 2004 Mar 29. PMID 15051639
- [Background] Cooper HA, Bloomfield DA, Bush DE, Katcher MS, Rawlins M, Sacco JD, Chandler M; AFFIRM Investigators. Relation between achieved heart rate and outcomes in patients with atrial fibrillation (from the Atrial Fibrillation Follow-up Investigation of Rhythm Management [AFFIRM] Study). Am J Cardiol. 2004 May 15;93(10):1247-53. doi: 10.1016/j.amjcard.2004.01.069. PMID 15135698
- [Background] Kaufman ES, Zimmermann PA, Wang T, Dennish GW 3rd, Barrell PD, Chandler ML, Greene HL; Atrial Fibrillation Follow-up Investigation of Rhythm Management investigators. Risk of proarrhythmic events in the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study: a multivariate analysis. J Am Coll Cardiol. 2004 Sep 15;44(6):1276-82. doi: 10.1016/j.jacc.2004.06.052. PMID 15364332
- [Background] Marshall DA, Levy AR, Vidaillet H, Fenwick E, Slee A, Blackhouse G, Greene HL, Wyse DG, Nichol G, O'Brien BJ; AFFIRM and CORE Investigators. Cost-effectiveness of rhythm versus rate control in atrial fibrillation. Ann Intern Med. 2004 Nov 2;141(9):653-61. doi: 10.7326/0003-4819-141-9-200411020-00005. PMID 15520421
- [Background] Shelton RJ. The AFFIRM study: approaches to control rate in atrial fibrillation. J Am Coll Cardiol. 2004 Dec 21;44(12):2418; author reply 2418-9. doi: 10.1016/j.jacc.2004.09.025. No abstract available. PMID 15607416
- [Background] Jenkins LS, Brodsky M, Schron E, Chung M, Rocco T Jr, Lader E, Constantine M, Sheppard R, Holmes D, Mateski D, Floden L, Prasun M, Greene HL, Shemanski L. Quality of life in atrial fibrillation: the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Am Heart J. 2005 Jan;149(1):112-20. doi: 10.1016/j.ahj.2004.03.065. PMID 15660042
- [Background] Olshansky B, Sami M, Rubin A, Kostis J, Shorofsky S, Slee A, Greene HL; NHLBI AFFIRM Investigators. Use of amiodarone for atrial fibrillation in patients with preexisting pulmonary disease in the AFFIRM study. Am J Cardiol. 2005 Feb 1;95(3):404-5. doi: 10.1016/j.amjcard.2004.09.044. PMID 15670555
- [Background] Cooper HA, Sacco J, Solomon AJ, Feld GK, Leman R, Wilber D; AFFIRM Investigators. Relation of initial resting ventricular rate to the ability to achieve and maintain normal sinus rhythm in patients with atrial fibrillation. Am J Cardiol. 2005 Mar 1;95(5):597-602. doi: 10.1016/j.amjcard.2004.10.037. PMID 15721098
- [Background] Curtis AB, Seals AA, Safford RE, Slater W, Tullo NG, Vidaillet H, Wilber DJ, Slee A. Clinical factors associated with abandonment of a rate-control or a rhythm-control strategy for the management of atrial fibrillation in the AFFIRM study. Am Heart J. 2005 Feb;149(2):304-8. doi: 10.1016/j.ahj.2004.08.012. PMID 15846269
- [Background] Murray KT, Rottman JN, Arbogast PG, Shemanski L, Primm RK, Campbell WB, Solomon AJ, Olgin JE, Wilson MJ, Dimarco JP, Beckman KJ, Dennish G, Naccarelli GV, Ray WA; AFFIRM Investigators. Inhibition of angiotensin II signaling and recurrence of atrial fibrillation in AFFIRM. Heart Rhythm. 2004 Dec;1(6):669-75. doi: 10.1016/j.hrthm.2004.08.008. PMID 15851238
- [Background] Wyse DG, Slee A, Epstein AE, Gersh BJ, Rocco T Jr, Vidaillet H, Volgman A, Weiss R, Shemanski L, Greene HL; AFFIRM Investigators. Alternative endpoints for mortality in studies of patients with atrial fibrillation: the AFFIRM study experience. Heart Rhythm. 2004 Nov;1(5):531-7. doi: 10.1016/j.hrthm.2004.07.007. PMID 15851214
- [Background] Sherman DG, Kim SG, Boop BS, Corley SD, Dimarco JP, Hart RG, Haywood LJ, Hoyte K, Kaufman ES, Kim MH, Nasco E, Waldo AL; National Heart, Lung, and Blood Institute AFFIRM Investigators. Occurrence and characteristics of stroke events in the Atrial Fibrillation Follow-up Investigation of Sinus Rhythm Management (AFFIRM) study. Arch Intern Med. 2005 May 23;165(10):1185-91. doi: 10.1001/archinte.165.10.1185. PMID 15911734
- [Background] Olshansky B, Heller EN, Mitchell LB, Chandler M, Slater W, Green M, Brodsky M, Barrell P, Greene HL. Are transthoracic echocardiographic parameters associated with atrial fibrillation recurrence or stroke? Results from the Atrial Fibrillation Follow-Up Investigation of Rhythm Management (AFFIRM) study. J Am Coll Cardiol. 2005 Jun 21;45(12):2026-33. doi: 10.1016/j.jacc.2005.03.020. PMID 15963405
- [Background] DiMarco JP, Flaker G, Waldo AL, Corley SD, Greene HL, Safford RE, Rosenfeld LE, Mitrani G, Nemeth M; AFFIRM Investigators. Factors affecting bleeding risk during anticoagulant therapy in patients with atrial fibrillation: observations from the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Am Heart J. 2005 Apr;149(4):650-6. doi: 10.1016/j.ahj.2004.11.015. PMID 15990748
- [Background] Flaker GC, Belew K, Beckman K, Vidaillet H, Kron J, Safford R, Mickel M, Barrell P; AFFIRM Investigators. Asymptomatic atrial fibrillation: demographic features and prognostic information from the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Am Heart J. 2005 Apr;149(4):657-63. doi: 10.1016/j.ahj.2004.06.032. PMID 15990749
- [Background] Curtis AB, Gersh BJ, Corley SD, DiMarco JP, Domanski MJ, Geller N, Greene HL, Kellen JC, Mickel M, Nelson JD, Rosenberg Y, Schron E, Shemanski L, Waldo AL, Wyse DG; AFFIRM Investigators. Clinical factors that influence response to treatment strategies in atrial fibrillation: the Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study. Am Heart J. 2005 Apr;149(4):645-9. doi: 10.1016/j.ahj.2004.09.038. PMID 15990747
- [Background] Olshansky B, Rosenfeld LE, Warner AL, Solomon AJ, O'Neill G, Sharma A, Platia E, Feld GK, Akiyama T, Brodsky MA, Greene HL; AFFIRM Investigators. The Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) study: approaches to control rate in atrial fibrillation. J Am Coll Cardiol. 2004 Apr 7;43(7):1201-8. doi: 10.1016/j.jacc.2003.11.032. PMID 15063430
- [Background] Chung MK, Shemanski L, Sherman DG, Greene HL, Hogan DB, Kellen JC, Kim SG, Martin LW, Rosenberg Y, Wyse DG; AFFIRM Investigators. Functional status in rate- versus rhythm-control strategies for atrial fibrillation: results of the Atrial Fibrillation Follow-Up Investigation of Rhythm Management (AFFIRM) Functional Status Substudy. J Am Coll Cardiol. 2005 Nov 15;46(10):1891-9. doi: 10.1016/j.jacc.2005.07.040. Epub 2005 Oct 21. PMID 16286177
- [Derived] Proietti M, Romiti GF, Olshansky B, Lip GYH. Systolic Blood Pressure Visit-to-Visit Variability and Major Adverse Outcomes in Atrial Fibrillation: The AFFIRM Study (Atrial Fibrillation Follow-Up Investigation of Rhythm Management). Hypertension. 2017 Nov;70(5):949-958. doi: 10.1161/HYPERTENSIONAHA.117.10106. Epub 2017 Oct 3. PMID 28974568
- [Derived] Saksena S, Slee A, Waldo AL, Freemantle N, Reynolds M, Rosenberg Y, Rathod S, Grant S, Thomas E, Wyse DG. Cardiovascular outcomes in the AFFIRM Trial (Atrial Fibrillation Follow-Up Investigation of Rhythm Management). An assessment of individual antiarrhythmic drug therapies compared with rate control with propensity score-matched analyses. J Am Coll Cardiol. 2011 Nov 1;58(19):1975-85. doi: 10.1016/j.jacc.2011.07.036. PMID 22032709
- Available data/document: Individual Participant Data Set: AFFIRM — http://biolincc.nhlbi.nih.gov/studies/affirm/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/affirm/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/affirm/